CLINICAL TRIAL: NCT01068119
Title: Feasibility and Safety of Same-Day Discharge of Troponin Negative Patients After Coronary PTCA Via the Transfemoral Approach
Brief Title: Same-Day Discharge After Coronary Percutaneous Transluminal Coronary Angioplasty (PTCA)
Acronym: GREECE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment and high number of screen failures
Sponsor: Piedmont Healthcare (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Dimitrios Karmpaliotis, MD, PhD, Piedmont Heart Institute/Piedmont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GREECE
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; percutaneous coronary angioplasty; Troponin negative; cardiac
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Same-day discharge (Experimental): Same-day discharge following PCI
  Interventions: Procedure: Same-day discharge

INTERVENTIONS:
Procedure: Same-day discharge — Patients identified as clinically stable are discharged home the same day as the PCI procedure with telephone follow-up at 12 hr, 24 hr, 3, 30, 180 and 365 days post procedure.

SUMMARY:
Same day discharge is safe and feasible in selected troponin negative patients undergoing coronary planned percutaneous coronary intervention (PCI) or ad hoc PCI via the transfemoral approach.

DETAILED DESCRIPTION:
The feasibility and safety of same day discharge post PCI will be examined. Study data will be compared to national registries and national or regional databases of PCI in Troponin negative patients with overnight stay. As part of the registry we will also assess compliance with dual antiplatelet therapy at six months and at 1 year and will record any reasons for premature discontinuation as well as any associated adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for catheterization/coronary angiography
2. Undergoing diagnostic coronary angiography to define the coronary anatomy with the intent for revascularization (ad-hoc PCI) or planned PCI to define the coronary anatomy with the intent for revascularization due to one of the following:

   1. exertional or rest chest pain (or angina equivalent)
   2. abnormal Exercise Stress Test
   3. abnormal nuclear tests
   4. abnormal pharmacologic or stress echocardiogram, or pharmacologic MRI
   5. abnormal EKGs
   6. abnormal Calcium scores
   7. abnormal coronary CT angiogram
3. Ability and willingness to consent and Authorization for use of PHI

Exclusion Criteria:

1. ACS (STEMI, UA/NSTEMI)
2. Positive Troponin I per local laboratory standards
3. Known EF<30%
4. GFR<50% (calculation using the IDMS-Traceable MDRD study equation
5. Dye Allergy that unable to be safely premedicated
6. Known current or history of bleeding diathesis
7. Current or anticipated treatment with warfarin, oral factor Xa inhibitor, oral direct thrombin inhibitor, LMWH, or TNK
8. Known platelet count <100,000/mm³ or known INR >1.5 at time of enrollment
9. Hgb <10 g/dL and/or Hct < 30%
10. Residence >60 minutes from the hospital
11. Reliable caregiver not available for home post PCI recovery
12. Participation in another study that would require hospital procedures or test post PCI prior to discharge
13. Inability or unwillingness to consent for study, follow up procedures and Authorization for use of PHI
14. Physician clinical determination participant is not suitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of cardiac MACE, major cerebral events, and groin complications | 6, 12, and 18 months post study initation

SECONDARY OUTCOMES:
Rate of compliance with dual antiplatelet therapy | 6, 12 , and 18 months post study initiation

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karmpaliotis, MD, PhD, Principal Investigator — Piedmont Heart Institute/Piedmont Hospital
Locations (1):
- Piedmont Hospital, Atlanta, Georgia, United States